CLINICAL TRIAL: NCT00431704
Title: Vinorelbine, Carboplatin and Trastuzumab in Advanced Her-2 Positive Breast Cancer, a Phase 2 Study
Brief Title: VinCaT: Vinorelbine, Carboplatin and Trastuzumab in Advanced Her-2 Positive Breast Cancer
Acronym: VinCaT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VinCaT; 2006-003994-28 (EudraCT Number)
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Metastatic Breast Cancer
Keywords: advanced; her-2 positive
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine; Carboplatin; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- vinorelbine, carboplatin, trastuzumab (Experimental)
  Interventions: Drug: vinorelbine; Drug: carboplatin; Drug: trastuzumab

INTERVENTIONS:
Drug: vinorelbine — 25 mg/m2 days 1 and 8 every 3 weeks for 6 cycles, or up to 9 cycles for responding patients
Drug: carboplatin — AUC 5 intravenously every 3 weeks for 6 cycles, up to 9 cycles for responding patients
Drug: trastuzumab — 8 mg/kg IV day 1, then 6 mg/kg IV every 3 weeks until disease progression

SUMMARY:
The purpose of this study is to evaluate the activity and safety of the combination of vinorelbine, carboplatin and trastuzumab in HER2-positive metastatic breast cancer.

DETAILED DESCRIPTION:
The addition of trastuzumab to chemotherapy containing anthracyclines or taxanes has improved survival in patients with Her-2 positive metastatic breast cancer, but newer combinations with less toxicity and cross resistance are needed. Early clinical studies have suggested that the combination of vinorelbine, carboplatin and trastuzumab can be active against metastatic breast cancer, with less toxicity. In this phase II single center trial, 39 patients will be enrolled to evaluate the activity and safety of this combination.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of breast cancer
* Stage IV disease
* None or at most one prior treatment for metastatic disease (prior treatment with trastuzumab for metastatic disease is not permitted)
* Overexpression of HER-2 (immunohistochemistry 3+) or genetic amplification of c-erbB2/neu (FISH+)
* ECOG Performance Status 0-2
* Age >18 and < 75 years
* Left Ventricular Ejection Fraction (LVEF) >50%
* Life expectancy >3 months
* Signed informed consent

Exclusion Criteria:

* Absence of measurable or evaluable disease
* Life expectancy < 3 months
* ECOG performance status > 2
* History of prior malignancy in the last 5 years (other than adequately treated non-melanoma skin cancer or excised cervical carcinoma in situ).
* Previous chemotherapy with vinorelbine or carboplatin (as adjuvant therapy or for metastatic disease)
* Previous therapy with trastuzumab for metastatic disease (previous adjuvant therapy with trastuzumab is permitted)
* Neutrophil < 2000/mm3, platelets < 100,000/mm3, haemoglobin < 9 g/dl
* Creatinine > 1.5 x the upper normal limits
* GOT and/or GPT > 2.5 x the upper normal limits and/or Bilirubin > 1.5 x the upper normal limits in absence of hepatic metastases
* GOT and/or GPT > 5 x the upper normal limits and/or Bilirubin > 3 x the upper normal limits in presence of hepatic metastases
* Congestive hearth failure or history of congestive heart failure, unstable angina pectoris even if it is medically controlled, myocardial infarction, clinically significant valve disease, uncontrolled arrhythmia
* Any concomitant pathology that would, in the investigator's opinion, contraindicate the use of the drugs in this study
* Male gender
* Pregnant or lactating women
* Refusal or incapacity to provide informed consent
* Inability to comply with follow up

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2007-10; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
objective response rate | after 3 and 6 cycles of therapy
side effects | after every cycle of therapy

SECONDARY OUTCOMES:
time to progression | at 12 months, end of study
overall survival | at 12 months, end of study

CONTACTS AND LOCATIONS:
Overall Officials: Andrea De Matteis, M.D., Principal Investigator — NCI Naples, Division of Medical Oncology C; Francesco Perrone, M.D., Ph.D., Principal Investigator — NCI Naples, Clinical Trials Unit
Locations (1):
- Istituto Nazionale dei Tumori, Divisione di Oncologia Medica C, Napoli, Italy